CLINICAL TRIAL: NCT03167814
Title: Prevention of Chyle-leak After Major Pancreatic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Tiina Vuorela, MD, PHd student, Junior surgeon, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUS/930/2017
Record Dates: First submitted 2017-05-15; First posted 2017-05-30 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Lymph Leakage; Chyle Into Mesentery; Extravasation; Pancreatic Cancer; Complication of Surgical Procedure
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients who fill our study ciriteria are asked to join in on the study and then they are randomized in to two groups, interventional and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet group (Active Comparator): Diet group will be on no-fat diet including MCT-oil supplement starting right after surgery according to our pancreas ERAS-protocol.
  Interventions: Dietary Supplement: Diet group
- Normal food-group (No Intervention): This study group will follow normal ERAS-protocol after pancreas surgery and start normal diet after surgery. If chyle-leak is diagnosed then it will be treated with the same no-fat diet as the intervention group.

INTERVENTIONS:
Dietary Supplement: Diet group — In the diet, there is no long-chain triglycerides. Fat and protein needs are met with adding medium-chain-fat acid as oil and protein supplements to the diet. Diet has been constructed together with clinical nutrition specialist.
  Arms: Diet group

SUMMARY:
Chyle is lymphatic fluid present in the wall of the intestine. It flows trough lymphatic vessels to cisterna chyli and to venous circulation carrying lymphatic fluid, long-chain triglyceride fatty acids and proteins, fatty soluble vitamins and electrolytes. Lymphatic vessels are at risk of damage in pancreatic surgery and especially when there is vein/artery resection and reconstruction at the same time. Chyle leak can be seen in post-operative patients when there is milky substance coming out of the surgical drains and drain fluids triglyceride level is high (>1,5 mmol/l). Patients with chyle leak are at risk of dehydration, malnutrition, sepsis and prolonged stay at the hospital. Usually treatment of chyle leak is with drains and no-fat diet up to 14 days after surgery. Sometimes combined with somatostatine-analogue-treatment. In this study investigators are randomizing patients with major pancreatic surgery in to two groups. Intervention group will start no-fat diet, including MCT-oil, right after surgery up to 2 weeks. And control group will start the diet if chyle-leak is seen. End goal is to reduce chyle-leaks in post-operative patients and analyze if it has an effect on patients prognosis.

DETAILED DESCRIPTION:
Patient who come for pancreatic surgery and vein resection/reconstruction will be randomized before surgery in two groups. Intervention group will start the no-fat diet right after surgery, with MCT-oil supplement. Diet will be continued up to 14 days after surgery. The control group will start the diet if chyle leak is diagnosed. Criteria of chyle leak in this study is appearance of milky-coloured fluid from the surgical drains in post-operative day 3 and drain fluids triglyceride levels must be high (>1,5 mmol/l). After enough patients have been recruited in the study, patient records are then analyzed to see if the no-fat diet has any effect on incidence of chyle-leak.

ELIGIBILITY:
Inclusion Criteria:

* Need for a pancreatic resection with vessel resection/reconstruction

Exclusion Criteria:

* No pancreatic and vessel resection needed
* Patients do not want to join the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Chyle-leakage reduced from operating area after surgery | 2 weeks after surgery or when patient is released from hospital, in the case of prolonged hospital-stay due to complications, is patient data being analyzed
  Post-operative chyle leak is diagnosed if drain fluids triglyserid content is above normal at post-operative day 3 (> 1,5mmol/l).

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Seppänen, Phd, Dos, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki university hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No